CLINICAL TRIAL: NCT03520439
Title: Mifepristone Versus Placebo to Treat Adenomyosis: a Double-blind, Multicentre，Randomized Clinical Trial
Brief Title: Evaluation of Therapeutic Effect and Safety of Mifepristone in the Treatment of Adenomyosis
Acronym: ETESRTA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: xinmei zhang (Other)
Collaborators: Anhui Province Cancer Hospital (Unknown); Huzhou Maternity and Child Care Hospital (Unknown); Jiaxing Maternity and Child Health Care Hospital (Other); Jinhua Municipal Central Hospital (Other); The Central Hospital of Lishui City (Other); The Affiliated Hospital of Medical School of Ningbo University (Unknown); Ningbo Maternity and Child Care Hospital (Unknown); The People's Hospital of Quzhou (Other); Shaoxing Women and Children's Hospital (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Taizhou First People's Hospital (Other); Zhoushan Maternity and Infant Hospital (Unknown); Shaoxing People's Hospital (Other)
Responsible Party: Sponsor-Investigator, xinmei zhang, Director, Women's Hospital School Of Medicine Zhejiang University
Organization: Women's Hospital School Of Medicine Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MF2018
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Adenomyosis
Keywords: Adenomyosis; mifepristone; the selective progesterone receptor modulators; treatment
MeSH Terms: conditions — Adenomyosis | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The appearance of Mifepristone Tablets and placebo tablets is the same (size, shape and color). In different treatment groups, the packaging of research drugs is the same, so that researchers or subjects or applicants can not know the assigned treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): mifepristone tablets ，10mg，One tablet daily, oral treatment
  Interventions: Drug: Mifepristone
- control group (Placebo Comparator): placebo，10mg，One tablet daily, oral treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mifepristone — Oral mifepristone 10mg (first menstrual third days), 1 times a day, 12 weeks, fasting or taking 2 hours after eating
  Other Names: RU486
  Arms: study group
Drug: Placebo — Oral Placebo Oral Tablet 1# (first menstrual third days), 1 times a day, 12 weeks, fasting or taking 2 hours after eating
  Arms: control group

SUMMARY:
This clinical trial is designed to study the effectiveness and safety of mifepristone in the treatment of symptomatic adenomyosis with multi center, random, double blind and controlled clinical trials. This multicenter study is performed in 150 subjects who are diagnosed as adenomyosis . Twelve weeks of randomization, allocation concealment, double-blind, placebo-controlled, parallel grouping. Subjects are randomly assigned to one of two treatment groups and received one of the following treatments:

1. Mifepristone tablets of 10mg, 1 tablet daily, oral
2. Placebo, 1 tablet daily, oral

DETAILED DESCRIPTION:
Adenomyosis is a common benign disease of Gynecology, with secondary progressive dysmenorrhea and menorrhagia as the main clinical manifestations, which seriously harm the physical and mental health of the patients. Most patients have the desire to retain the uterus. Therefore, the treatment of drug conservative treatment is dominant in the treatment of adenomyosis. However, the current clinical treatment of adenomyosis still has some limitations and needs to be improved. Therefore, it is imperative to expand the clinical medication of adenomyosis.

Mifepristone is defined as a selective progesterone receptor modulator. Under specific conditions, it plays the role of anti progestin, inhibits endometrial proliferation, inhibits ovulation, and can cause reversible amenorrhea. In recent years, it has been widely used in of uterine leiomyoma and endometriosis. Adenomyosis is also closely related to hormone related diseases, especially endometriosis. At present, the study of mifepristone in the treatment of adenomyosis is more extensive in China. A large number of domestic literature reports that low dose mifepristone for the treatment of adenomyosis is safe and effective for the treatment of adenomyosis . During the treatment of mifepristone, most of the patients had amenorrhea, obviously alleviating dysmenorrhea and reducing the menstrual volume, reducing the uterine and lesion volume of the patients with adenomyosis . However, most of the domestic literature is a small sample case control study or retrospective study. There is no randomized double blind control study. There is no clinical study on the application of mifepristone to adenomyosis in foreign countries. Therefore, the clinical evidence is inadequate, and a high quality randomized controlled trial is still needed. The purpose of this study is to demonstrate the effectiveness and safety of mifepristone (10mg) in the treatment of symptomatic adenomyosis with multi center, random, double blind and controlled clinical trials. It is a new clinical study for the old medicine.

ELIGIBILITY:
Inclusion Criteria:

1. B-ultrasound or magnetic resonance imaging (MRI) examination confirmed that the subject has adenomyosis, and the uterus is less than 10 weeks of pregnancy;
2. Visual analogue scale (VAS) of adenomyosis-associated pain> 0 points; with or without menorrhagia (PBAC≥100 points);
3. Women between 18 and 50 years old who currently have no childbearing requirements;
4. Normal or cervical cytology results without clinical significance (results within 6 months before the screening period);
5. Willing to choose a barrier method of contraception if contraception is needed;
6. Be tested voluntarily and sign the informed consent.
7. No menopause

No menopause

Exclusion Criteria:

1. HB<90G/L
2. Undiagnosed abnormal vaginal bleeding or endometrial lesions;
3. Pregnancy and lactation women and those who are preparing to give birth when taking the medication or within 6 months of stopping the medication;
4. Malignant tumors (including the reproductive system and other systems);
5. The patients with severe heart, liver, kidney disease and adrenocortical insufficiency;
6. The results of follow-up laboratory test indicate abnormal clinical significance;
7. The allergic persons or those who have been allergic to multiple drugs, or are allergic to active ingredients or any excipients of the study drug;
8. Suffering from any disease or condition that may cause the study drug to alter absorption, accumulate excessively, affect metabolism, or change the excretion pattern;
9. Having clinically significant depression within the current or most recent year;
10. People who regularly take analgesics due to other underlying diseases;
11. Ketoconazole, itraconazole, erythromycin, rifampicin, corticosteroids (hydrocortisone, prednisone, dexamethasone, etc.), and some anticonvulsants (phenytoin, phenobarbital, carbamazepine, etc.), griseofulvin, non-steroidal anti-inflammatory drugs (aspirin, acetaminophen, etc.) that are being used and cannot be stopped during the study;
12. Previous use of hormone drugs, including: a. use of GnRH agonists within 6 months before the screening period; b. use of progestins or danazol and other long-acting hormones within 3 months before the screening period; c. use of oral contraceptive-like short-acting hormones within one month before the screening period;
13. Patients who participated in other clinical trials within 3 months before the screening, or who are considered inappropriate to participate in the study by other investigators.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2018-05-19 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
changes in chronic pelvic pain associated with adenomyosis | Baseline ,taking medicine for 1-month, 2-month, 3-month and post treatment 1- month（approximately 16 weeks）
  To evaluate the visual analogue scale (VAS) changes.By using 10-cm visual analogue scales (0 = no pain, 10 = worst pain). Women will be asked to give the pain score at each follow up (i.e.Baseline ,taking medicine for 1-month, 2-month, 3-month, post treatment 1- month )

SECONDARY OUTCOMES:
changes in uterine bleeding | Baseline ,taking medicine for 1-month, 2-month, 3-month and post treatment 1- month（approximately 16 weeks）
  To evaluate the pictorial blood loss assessment chart (PBAC) changes
improvement of anemia | Baseline ,taking medicine for 1-month, 3-month （approximately 16 weeks）
  To evaluate the hemoglobin changes,
Size of uterus | Baseline ,taking medicine for 1-month, 3-month （approximately 16 weeks）
  To evaluate the uterine volume changes

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital of Zhejiang Medical University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Che X, Wang J, Sun W, He J, Wang Q, Zhu D, Zhu W, Zhang J, Dong J, Xu J, Zheng F, Zhou J, Zhao W, Lin Q, Ye L, Zhao X, Xu Z, Chen Y, Wang J, Wu W, Zhai L, Zhou Y, Zheng J, Zhang X. Effect of Mifepristone vs Placebo for Treatment of Adenomyosis With Pain Symptoms: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2317860. doi: 10.1001/jamanetworkopen.2023.17860. PMID 37307001